CLINICAL TRIAL: NCT02890576
Title: Organization of Ambulatory Telemonitoring of People With Hearing Loss and Having a Cochlear Implant.
Brief Title: Ambulatory Telemonitoring of People With Hearing Loss and Having a Cochlear Implant COCHLESURV
Acronym: COCHLESURV
Status: Withdrawn | Type: Observational
Why Stopped: study was stopped du to of patient lack
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 13 6900 15
Record Dates: First submitted 2016-07-21; First posted 2016-09-07 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Deafness
Keywords: cochlear implant; telemedicine; new organization of patient monitoring
MeSH Terms: conditions — Deafness | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- telemedicine: Setting up of a new organization of medical monitoring (ussing telemedicine) of patient having a cochlear implant
  Interventions: Other: telemedicine

INTERVENTIONS:
Other: telemedicine — Monitoring of patients with cochlear implant with sessions of telemedicine

SUMMARY:
The number of patients with cochlear implants increases every year, constituting an active queue increasingly important (60 new cases per year in Toulouse, active list in 2013: 380 adult patients). The number of approved cochlear implant centers is limited by guardianships, and corresponds to the Hospitals University. It is not possible to create networks of correspondents. Teams of implantation centers must meet the needs of new patients and ensure continuity of care for patients already implanted: speech therapy monitoring, adjustment and rehabilitation.

In case of malfunction of the implant, patients use in first-line reference center. The increasing number of patients leads to a lack of specialized teams that can not meet the demands of patients in a timely manner, while continuing to provide support for new patients. It is therefore necessary to find solutions to improve the service provided to patients who received a cochlear implant system to respond quickly and effectively to the request of troubled patients, while optimizing the workload of the teams . The introduction of a telemedicine platform is expected to achieve these goals, distinguishing minor malfunctions, not requiring a consultation in a center, and the most complex situations requiring consultation in a center.

DETAILED DESCRIPTION:
The strategy of the study is to establish contact with the patient at home in case of problems through the establishment of a daily continuously in service by telephone contact and video calling.

There will be no change in the usual care of the patient. The monitoring center by health professionals (speech therapists, technicians and doctors ORL) in the cochlear implant center will operate a daily permanence of 5 half days on business days, to respond to a patient call.

Are excluded from this research, emergency management such as meningitis, which passes through the usual emergency lane.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years), carrying a cochlear implant,
* Familiar with using the Internet and with equipment (computer and computer video camera) at his home
* Agreeing to participate in the study,
* With a social protection system.

Exclusion Criteria:

* Misunderstanding of login procedures,
* Failure to follow procedures,
* Person under a legal protection system (guardianship, curators or safeguard justice)
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with deafness and having a cochlear implant
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
the number of movements avoided the center, | 12 months after the inclusion
  number of contacts have avoided moving the patient to the center

SECONDARY OUTCOMES:
The delay for the identification of malfunction | Up to 1 year
The time spent by the health professional during a telemedicine session | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Deguine, MD, PhD, Principal Investigator — Hospital University of Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272